CLINICAL TRIAL: NCT07187830
Title: Region-specific Adipose Tissues and Liver Changes Associated With Semaglutide Treatment in Chronic Kidney Disease Patients
Brief Title: Visceral Adipose Tissue and Liver Changes Associated With Semaglutide in CKD
Acronym: ADIPOLIVE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Novo Nordisk Canada Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: U1111-1328-1600
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease in Type 2 Diabetes; Obesity & Overweight
Keywords: chronic kidney disease; cardiovascular disease; obesity; diabetes mellitus; steatosis
MeSH Terms: conditions — Obesity; Overweight; Renal Insufficiency, Chronic; Cardiovascular Diseases; Diabetes Mellitus; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Urine, blood and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- No semaglutide: Patients with diabetes not treated with semaglutide
- Semaglutide: Patients with diabetes receiving semaglutide

SUMMARY:
Obesity is considered a global pandemic and is associated with various diseases and metabolic complications, such as type 2 diabetes mellitus, high blood pressure, cholesterol disorders, cancer, cardiovascular disease, and kidney disease. Obesity can affect the kidneys in two main ways: indirectly, through mechanisms related to diabetes mellitus and/or high blood pressure, and directly, through complex proteins called "adipokines," which are produced by adipocytes.

Many of these adipokines are secreted by adipocytes under normal conditions, as they contribute to maintaining immune defenses and energy production. However, in obesity these adipokines acquire harmful properties and produce chronic inflammation in vital organs, such as the heart, blood vessels, the pancreas, and the kidney, leading to a deterioration in liver and kidney function.

New drugs such as glucagon-like peptide-1 receptor agonists (GLP-1Ras / Semaglutide), are not only effective to regulate blood sugar levels, but they produce weight loss improving kidney and liver function. However, little is known about their specific effect on the adipose tissue. Therefore, studies focusing on how these drugs work in fat could help us understand how diseased adipose tissue can affect patients with heart, liver, and kidney disease.

Investigators are asking patients who attend the diabetes clinics associated with the University of Alberta to join the study.

DETAILED DESCRIPTION:
If participants agree to join the study, they will be asked to undergo a magnetic resonance imaging (MRI) scan to measure the fat around the heart, liver, and kidneys. During the abdominal MRI scan, the fat content of the liver will also be measured.

When participants arrive for the imaging test, they will first sign an informed consent form. Participants will then proceed to have their MRI imaging test.

The MRI imaging study will be performed in the MRI Research Center on the lower level of the Mazankowski Alberta Heart Institute (part of the University Hospital). Study personnel will also ask participants questions about their medical history. Other information collected will include medications, recent tests the participants' doctor may have ordered, and basic information such as age, sex, weight, and height.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age.
* Patients diagnosed with T2DM (>18 months) and CKD in stages G1, G2, G3a, G3b and G4; the CKD staging will be established according to the eGFR as per the KDIGO guidelines (G1: eGFR ≥90 ml/min/1.73m2; G2: 60-89 ml/min/1.73m2; G3a: 45-59 ml/min/1.73m2; G3b: 30-44 ml/ min/1.73m2; G4: 15-29 ml/ min/1.73m2).
* Patients with T2DM and CKD, with or without semaglutide treatment.
* Patients who voluntarily agree to participate and sign informed consent.

Exclusion Criteria:

* Patients <18 years of age.
* Pregnant, breastfeeding, or an intention of becoming pregnant or not using adequate contraceptive measures (including country-specific adequate measures, if any)
* Patients diagnosed with T2DM and CKD in stage G5 or stage G4 requiring dialysis as per KDIGO guidelines.
* Previous participation in this trial (screened or randomized)
* Patients diagnosed with neuropsychiatric diseases that prevent them from understanding the benefits/risks associated with the project or voluntarily choosing to participate.
* Known or suspected allergy to trial medication(s), excipients, or related products
* Contraindications to study medication(s), worded specifically as stated in the Product Monograph
* Refusal to participate or consent revocation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll patients with diabetic kidney disease at different stages of CKD receiving the GLP-1RA Semaglutide or SoC regimen, depending on their medical indication and cardiometabolic and hepatic steatosis stage.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between kidney disease progression and cardiometabolic changes | From enrollment to the end of follow-up at 12 months
  To establish a correlation between kidney disease progression and cardiometabolic changes, focusing on region-specific adipose tissues such as perirenal, epicardial, and hepatic steatosis in patients with or without semaglutide treatment.

SECONDARY OUTCOMES:
Adiposopathy biomarkers in different CKD stages | From enrollment to the end of follow-up at 12 months
  Adiposopathy biomarker comparisons between different CKD severity stages will be investigated

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Raggi, M.D, Principal Investigator — University of Alberta; Luis G D'Marco, M.D; Ph,D., Principal Investigator — CEU Cardenal Herrera University
Locations (1):
- Mazankowski Alberta Heart Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT07187830/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT07187830/ICF_001.pdf